CLINICAL TRIAL: NCT02891161
Title: Phase Ib/II Study of Concurrent Durvalumab And Radiation Therapy (DUART) Followed by Adjuvant Durvalumab in Patients With Urothelial Cancer (T2-4 N0-2 M0) of the Bladder: Big Ten Cancer Research Consortium BTCRC-GU15-023
Brief Title: Durvalumab And Radiation Therapy Followed by Adjuvant Durvalumab in Patients With Urothelial Cancer (T2-4 N0-2 M0) of the Bladder
Acronym: DUART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor-investigator elected to discontinue followup on remaining subjects after planned analyses and manuscripts were completed.
Sponsor: Monika Joshi, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Monika Joshi, MD, M.D., Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GU15-023
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Urothelial Cancer
Keywords: durvalumab; MEDI4736; anti-PD-L1
MeSH Terms: interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Safety Run In Phase Ib (Experimental): Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  Interventions: Drug: durvalumab; Radiation: Radiation Therapy
- Arm B: Investigational Treatment Phase II (Experimental): Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2.. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Adjuvant durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  Interventions: Drug: durvalumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: durvalumab — 1500 mg Q4 weekly
Radiation: Radiation Therapy — 64.8 Gy, 36 daily fractions on weekdays over about 7 weeks
  Other Names: RT

SUMMARY:
This is an open label, multi-institutional, single arm study of a phase Ib study, followed by a phase II study of durvalumab with radiation therapy (RT) in patients with urothelial cancer (UC). No randomization or blinding is involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

The phase Ib study will evaluate the safety of combining durvalumab with RT followed by adjuvant durvalumab. The phase II study will estimate the Progression Free Survival (PFS) and Disease Control Rate (DCR) with durvalumab plus RT followed by single agent durvalumab for patients with UC of bladder.

PHASE Ib INVESTIGATIONAL TREATMENT:

Cohort 1 will consist of up to 6 patients who will receive durvalumab 1500mg 2 doses Q4 weekly with RT to gross disease, 64.8 Gy, 36 fractions on weekdays over about 7 weeks. Durvalumab will be started on day 1; RT will be started on day 1 or 2.

Three patients will be enrolled initially. If 2 or more patients (out of 3) experience dose-limiting toxicity (DLT), the combined treatment will be considered unsafe. Otherwise, an additional 3 patients will be treated at the same dose. If 0 or 1 patient experience DLT, the dose of durvalumab will be deemed safe for phase 2 part of the study. If, however, 2 or more patients (out of 6) experience DLT, the combined treatment will be considered unsafe.

Post-concurrent durvalumab and RT, single agent durvalumab will be given1500mg every 4 weeks (±7 days) for a total period of up to 12 months. Adjuvant durvalumab treatment will be started 3-4 weeks post completion of durvalumab and RT.

PHASE II INVESTIGATIONAL TREATMENT:

Subjects will receive durvalumab 1500mg 2 doses Q4 weekly with RT to gross disease, 64.8 Gy, 36 fractions on weekdays over about 7 weeks. Durvalumab will start on Day 1. RT to start on Day 1 or 2.

Post-concurrent durvalumab and RT, single agent durvalumab will be given1500mg every 4 weeks (±7 days) for a total period of up to 12 months. Adjuvant durvalumab monotherapy will be started 3-4 weeks post completion of durvalumab and RT.

Life expectancy of >6 months per treating physician.

Adequate organ and marrow function as defined below:

1. Hemoglobin ≥ 9.0 g/dL
2. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
3. Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3)
4. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN.
6. Serum creatinine CL>30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

ELIGIBILITY:
Inclusion Criteria:

Phase Ib subjects must meet the following inclusion criteria:

* Locally advanced urothelial cancer of bladder with any of the following:

  1. T3-4, N0-2 M0, OR Tx N1-2 M0 OR T2 N1-2 M0: Treatment naïve, unresectable, OR medically unfit for surgery, OR cisplatin ineligible. T3 N0 M0 patients can be included if they are cisplatin ineligible.
  2. Patients who have T3-4, N0-2 M0 OR Tx N1-2 M0 OR T2 N1-2 M0 post-neoadjuvant chemotherapy who become unresectable OR medically unfit for surgery.

     Phase II subjects must meet the following inclusion criteria:
* Locally advanced urothelial cancer of bladder with any of the following:

  1. T3-4, N0-2 M0 OR Tx N1-2 M0 OR T2 N1-2 M0: Treatment naïve, unresectable, OR medically unfit for surgery OR cisplatin ineligible. T3 N0 M0 patients can be included if they are cisplatin ineligible.
  2. T3-4, N0-1 M0 OR Tx N1-2 M0 OR T2 N1-2 M0 patients post-neoadjuvant chemotherapy who become unresectable OR medically unfit for surgery.
* T2, N0, M0 who are ineligible to get cisplatin based chemotherapy.

All subjects:

* Written informed consent and HIPAA authorization for personal health information, obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy of >6 months per treating physician.
* Subjects must have archival tissue available from previous TURBT (preferred) or lymph node core biopsy within 8 weeks of treatment or be assessed by the treating urologist to undergo maximal TURBT. The extent of TURBT may vary for each patient and will be determined by the treating urologist. Further, the treating urologist will decide if performing the TURBT is clinically appropriate. If the potential subject does not have tumor amenable to biopsy, there is insufficient tissue for PD-L1 testing or is not clinically appropriate for TURBT, enrollment must be discussed with the sponsor-investigator on a case by case basis.
* Histologically proven urothelial carcinoma of bladder with predominant transitional cell component. Adenocarcinoma, squamous cell differentiation, or other atypical histology (such as plasmacytoid or sarcomotoid) of the bladder will be allowed on the study, provided they form <50% of the histology
* Females of childbearing potential must have a negative urine and serum pregnancy test within 3 days of study registration.

NOTE: Female subjects are considered of child bearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are ≥60 years old and naturally postmenopausal for at least 12 consecutive months.

* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Participation in another clinical study with an investigational product within 2 weeks prior to registration.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
* Previous systemic immunotherapy. Previous use of intravesical BCG is acceptable.
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence. However adequately treated prostate cancer >3 years ago with no significant change in PSA for past 6 months can be included. Patients with a history of prostate cancer must not have any definitive radiation therapy to prostate area.
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within14 days prior to the first dose of study drug (14 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms on electrocardiogram (ECG) using Frediricia's Correction.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy. (Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy).
* Any prior Grade ≥3 Immune-mediated adverse event (imAE) while receiving any previous immunotherapy agent, or any unresolved imAE >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with h/o completely resolved childhood asthma or atopy will not be excluded. Patients with well-controlled hypothyroidism on thyroxine replacement will be eligible as well.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of and/or confirmed pneumonitis.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to durvalumab or any excipient.
* History of hypersensitivity to the combination or radiation therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known history of previous clinical diagnosis of tuberculosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of starting treatment with durvalumab.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control. For this study male or female patients of reproductive potential need to employ two highly effective and acceptable forms of contraception throughout their participation in the study and for 90 days after last dose of study drug
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Brain metastases or history of leptomeningeal carcinomatosis.
* Subjects with uncontrolled seizures.
* Previous definitive radiation to pelvic area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, MD, MRCP, Principal Investigator — Penn State Cancer Institute
Locations (7):
- United States (7):
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Penn State Cancer Intsitute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert & The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Joshi M, Tuanquin L, Zhu J, Walter V, Schell T, Kaag M, Kilari D, Liao J, Holder SL, Emamekhoo H, Sankin A, Merrill S, Zheng H, Warrick J, Hauke R, Gartrel B, Stein M, Drabick J, Degraff DJ, Zakharia Y. Concurrent durvalumab and radiation therapy (DUART) followed by adjuvant durvalumab in patients with localized urothelial cancer of bladder: results from phase II study, BTCRC-GU15-023. J Immunother Cancer. 2023 Feb;11(2):e006551. doi: 10.1136/jitc-2022-006551. PMID 36822667
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm Ib: Safety Run In Phase Ib: Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
  Radiation Therapy: 64.8 Gy, 36 daily fractions on weekdays over about 7 weeks
- Arm II: Investigational Treatment Phase II: Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Adjuvant durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
Period: Study Treatment
Arm/Group | Arm Ib: Safety Run In Phase Ib | Arm II: Investigational Treatment Phase II
Started | 6 | 20
Completed | 2 | 7
Not Completed | 4 | 13
Not completed — Disease Progression | 2 | 4
Not completed — AE/Side Effects/Complications | 1 | 5
Not completed — Patient withdrawal After Therapy Start | 1 | 4
Period: Follow up
Arm/Group | Arm Ib: Safety Run In Phase Ib | Arm II: Investigational Treatment Phase II
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 6 | 20
Completed | 2 | 3
Not Completed | 4 | 17
Not completed — Death | 4 | 8
Not completed — Refused to Follow up | 0 | 2
Not completed — Symptomatic deterioration | 0 | 1
Not completed — Study terminated | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm Ib: Safety Run In Phase Ib | Arm II: Investigational Treatment Phase II | Total
Number analyzed (Participants) | 6 | 20 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (14.05) | 76.6 (7.44) | 75 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 5 | 14 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 18 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 1 | 1
  Ethnicity: Non-Hispanic | 5 | 18 | 23
  Ethnicity: Unknown | 1 | 1 | 2
Tumor Node Metastasis (TNM) stage at screening [Count of Participants; unit: Participants] — Primary tumor (T) TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4:The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Regional lymph nodes (N) NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: The higher the number after the N, the more lymph nodes that contain cancer.
  Distant metastasis (M) MX: Metastasis cannot be measured. M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    T2N0M0 | 0 | 10 | 10
    T2N1M0 | 1 | 2 | 3
    T2N2M0 | 0 | 1 | 1
    T3N0M0 | 1 | 5 | 6
    T3N2M0 | 1 | 1 | 2
    T4N0M0 | 1 | 0 | 1
    T4N1M0 | 1 | 0 | 1
    T4N2M0 | 1 | 0 | 1
    T4NXMX | 0 | 1 | 1
Unresectable [Count of Participants; unit: Participants]
  Subject's tumor is unresectable at screening. | 3 | 6 | 9
  Subject's tumor is not unresectable at screening. | 3 | 14 | 17
Unfit for surgery [Count of Participants; unit: Participants]
  Subject is medically unfit for surgery at screening | 2 | 11 | 13
  Subject is not medically unfit for surgery at screening | 4 | 9 | 13
Cisplatin ineligible [Count of Participants; unit: Participants]
  Subject is cisplatin ineligible at screening | 4 | 19 | 23
  Subject is not cisplatin ineligible at screening | 2 | 1 | 3
ECOG status [Count of Participants; unit: Participants] — 0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0-1 | 5 | 14 | 19
    2 | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Safety Assessment - Evaluation of DLT (Dose Limiting Toxicity) Rate
Description: To assess the safety of combining durvalumab with RT in that DLT rate is lower than than 33% based on CTCAEv4.0
Time Frame: Begin W1 and every 2 chemotherapy cycles (2 weeks) thereafter, for up to 2 years or until unacceptable toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Ib: Safety Run In Phase Ib
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: All Phases: Progression Free Survival Rate at 1 Year
Description: Progression free survival rate at one year is defined as the probability that a patient remains free of progression of disease (SD+CR+PR) by modified RECIST 1.1 and cystoscopy at 1 year from the start of durvalumab treatment, D1 of durvaRT.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From C1D1 to Progression or until death for 1 year
Population: All Phase Ib and Phase II subjects were analyzed together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase Ib and II: Arm Ib: Safety Run In Phase Ib Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
  Radiation Therapy: 64.8 Gy, 36 daily fractions on weekdays over about 7 weeks
  Arm II: Investigational Treatment Phase II
  Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Adjuvant durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
Arm/Group | Phase Ib and II
Number analyzed (Participants) | 26
percentage of participants | 71.5 [55.6 to 91.9]

3. Primary Outcome: Phase II: Disease Control Rate to Concurrent durvaRT Followed by Durvalumab
Description: The number of all subjects is reported with stable disease (SD) for 8 weeks, or partial response (PR), or complete response (CR) according to modified RECIST 1.1 and cystoscopy, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease(SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started;Disease Control Rate (DCR) = CR + PR+SD
Time Frame: From C1D1 until death or up to a maximum of 39 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II: Investigational Treatment Phase II
Number analyzed (Participants) | 20
Participants | 13

4. Secondary Outcome: All Phases: DCR Post Completion of Concurrent durvaRT
Description: We will be determining the disease control rate, defined as percentage of patients achieving CR, PR, SD post completion of concurrent durvaRT. This will give us some preliminary evidence for efficacy of durvaRT combination.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease(SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started;Disease Control Rate (DCR) = CR + PR+SD
Time Frame: From C1D1 until death or up to a maximum of 39 months
Population: Phase Ib and Phase II subjects were analyzed together.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase Ib and Phase II: Arm Ib: Safety Run In Phase Ib Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
  Radiation Therapy: 64.8 Gy, 36 daily fractions on weekdays over about 7 weeks
  Arm II: Investigational Treatment Phase II
  Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Adjuvant durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
Arm/Group | Phase Ib and Phase II
Number analyzed (Participants) | 26
percentage of participants | 72.7 [51.8 to 86.8]

5. Secondary Outcome: All Phases : Median Progression Free Survival (PFS) Time
Description: Median progression free survival will be determined for all subjects.
Time Frame: From C1D1 to PD or until death or up to a maximum of 37 months.
Population: Phase Ib and Phase II subjects were analyzed together
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Phases: Arm Ib: Safety Run In Phase Ib Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
  Radiation Therapy: 64.8 Gy, 36 daily fractions on weekdays over about 7 weeks
  Arm II: Investigational Treatment Phase II
  Subjects will receive durvalumab 1500mg Q4 weekly with RT to gross disease over 36 fractions. Durvalumab will start on Day 1. RT to start on Day 1 or 2. Subjects will receive adjuvant durvalumab monotherapy Q4 week, up to 12 months. Adjuvant durvalumab monotherapy to start 4 weeks post completion of durvalumab and RT.
  durvalumab: 1500 mg Q4 weekly
Arm/Group | All Phases
Number analyzed (Participants) | 26
months | 21.8 [14.8 to NA] — upper limit was not reached due to insufficient number of participants with events.

6. Secondary Outcome: Phase II: Complete Remission
Description: Estimate the rate of CR is one of the secondary objectives for phase II part of this study. This will help us determine the actual effectiveness of durvaRT approach. CR will be determined with the help of imaging and cystoscopy post completion of durvaRT per modified RECIST 1.1.
  Number of subjects reporting CR will be reported here. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions.
Time Frame: From C1D1 until CR or death or up to a maximum of 39 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II: Investigational Treatment Phase II
Number analyzed (Participants) | 20
Participants | 17

7. Secondary Outcome: All Phases: Overall Survival
Description: Estimate the overall survival (OS), defined as time from start of treatment, D1, to the date of death due to any cause. OS is defined, as time from start of treatment to the date of death due to any cause, or to the date of censoring at the last time the subject was known to be alive in intention-to-treat population. OS is one of the secondary objectives of this study. This is an immunotherapy based clinical trial and it is prudent to determine the OS to reflect the long-term benefit from this therapeutic approach.
Time Frame: From C1D1 until death or 39 months.
Population: Phase Ib and Phase II subjects were analyzed together.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Phases
Number analyzed (Participants) | 26
months | 30.8 [21.8 to NA] — upper limit was not reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from week 1 of treatment and every 2 chemotherapy cycles (2 weeks) thereafter, for up to 39 months or until unacceptable toxicity. All-Cause Mortality was assessed from week 1 of treatment and every 2 chemotherapy cycles (2 weeks) thereafter, for up to 39 months or until unacceptable toxicity
Description: An Adverse Event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Arm Ib: Safety Run In Phase Ib | Arm II: Investigational Treatment Phase II
All-Cause Mortality (participants affected / at risk) | 4/6 | 8/20
Serious Adverse Events (participants affected / at risk) | 4/6 | 8/20
Other Adverse Events (participants affected / at risk) | 6/6 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Ib: Safety Run In Phase Ib (N=6) | Arm II: Investigational Treatment Phase II (N=20)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
STROKE (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 0 (0) | 1 (2)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 0 (0) | 1 (4)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (3)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Ib: Safety Run In Phase Ib (N=6) | Arm II: Investigational Treatment Phase II (N=20)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (5) | 4 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (4)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
ANEMIA (Blood and lymphatic system disorders) | 6 (10) | 10 (12)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
ANXIETY (Psychiatric disorders) | 2 (2) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 3 (4)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
BRUISING (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
CARDIAC DISORDERS (Cardiac disorders) | 2 (4) | 6 (10)
CHOLESTEROL HIGH (Investigations) | 1 (1) | 7 (7)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 12 (14)
CREATININE INCREASED (Investigations) | 3 (8) | 13 (17)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 3 (5) | 6 (8)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2) | 4 (7)
DEPRESSION (Psychiatric disorders) | 2 (2) | 4 (4)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (2) | 12 (23)
DIZZINESS (Nervous system disorders) | 1 (1) | 6 (7)
DRY EYE (Eye disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
EDEMA LIMBS (General disorders) | 3 (6) | 11 (16)
ENDOCRINE DISORDERS (Endocrine disorders) | 2 (2) | 4 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 5 (9) | 15 (21)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 11 (13)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 4 (4) | 6 (8)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
GGT INCREASED (Investigations) | 2 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 4 (4)
HEARING IMPAIRED (Ear and labyrinth disorders) | 2 (2) | 3 (3)
HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 3 (6) | 10 (16)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (5) | 3 (4)
HYPERKALEMIA (Metabolism and nutrition disorders) | 3 (3) | 7 (22)
HYPERTENSION (Vascular disorders) | 3 (3) | 17 (45)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERURICEMIA (Metabolism and nutrition disorders) | 2 (3) | 8 (15)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (4) | 4 (8)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (3) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 3 (3)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 2 (2) | 4 (5)
INFUSION RELATED REACTION (General disorders) | 1 (1) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
INSOMNIA (Psychiatric disorders) | 1 (1) | 5 (6)
INVESTIGATIONS (Investigations) | 1 (1) | 5 (6)
LARYNGEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (22) | 8 (19)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 2 (4) | 4 (6)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (6)
NAIL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (5) | 5 (10)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (3) | 3 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (9)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 3 (5) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
PROTEINURIA (Renal and urinary disorders) | 1 (2) | 2 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6)
RECTAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 4 (6) | 11 (18)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 1 (1) | 4 (4)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
SERUM AMYLASE INCREASED (Investigations) | 1 (1) | 5 (7)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 3 (7) | 6 (9)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 2 (2)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
TRIGEMINAL NERVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 4 (5) | 5 (5)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 4 (9) | 11 (29)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 3 (3)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 7 (8)
URINARY URGENCY (Renal and urinary disorders) | 3 (3) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
VASCULAR DISORDERS (Vascular disorders) | 1 (1) | 3 (4)
VOMITING (Gastrointestinal disorders) | 2 (3) | 4 (8)
WEIGHT LOSS (Investigations) | 2 (2) | 3 (7)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (13) | 3 (3)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 4 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 1 (2)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 4 (4)
BLURRED VISION (Eye disorders) | 0 (0) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC TROPONIN T INCREASED (Investigations) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 4 (5)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 8 (8)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (3)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
EYE DISORDERS (Eye disorders) | 0 (0) | 6 (10)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 5 (7)
FEVER (General disorders) | 0 (0) | 4 (7)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (2)
FLOATERS (Eye disorders) | 0 (0) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 0 (0) | 1 (1)
GENITAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 2 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 2 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 5 (6)
INR INCREASED (Investigations) | 0 (0) | 1 (1)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LIPASE INCREASED (Investigations) | 0 (0) | 4 (16)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
MOBITZ (TYPE) II ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 4 (4)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 2 (2)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
SCLERAL DISORDER (Eye disorders) | 0 (0) | 1 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 3 (5)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
STOMAL ULCER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 3 (3)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 4 (4)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 3 (3)
URINE DISCOLORATION (Renal and urinary disorders) | 0 (0) | 1 (2)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VITREOUS HEMORRHAGE (Eye disorders) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 0 (0) | 3 (4)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT02891161/Prot_SAP_000.pdf